CLINICAL TRIAL: NCT06132893
Title: A Phase 2/3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Efficacy, Safety and Tolerability of BHV-7000 in Subjects With Refractory Focal Onset Epilepsy
Brief Title: A Study to Determine if BHV-7000 is Effective and Safe in Adults With Refractory Focal Onset Epilepsy
Acronym: RISE 2
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV7000-302; 2023-508539-30 (Registry Identifier: EU CTR)
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Focal Epilepsy
Keywords: Focal Epilepsy; Epilepsy; Seizure; Refractory Epilepsy; Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures; Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BHV-7000 25 mg Part A (Experimental)
  Interventions: Drug: BHV-7000
- BHV-7000 50 mg Part A (Experimental)
  Interventions: Drug: BHV-7000
- Placebo Part A (Placebo Comparator)
  Interventions: Drug: Placebo
- BHV-7000 75 mg Part B (Experimental)
  Interventions: Drug: BHV-7000
- Placebo Part B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 25 mg. Participants will take blinded investigational product (IP) once daily
  Arms: BHV-7000 25 mg Part A
Drug: BHV-7000 — BHV-7000 50 mg. Participants will take blinded investigational product (IP) once daily
  Arms: BHV-7000 50 mg Part A
Drug: Placebo — Matching placebo taken once daily
  Arms: Placebo Part A
Drug: BHV-7000 — BHV-7000 75 mg. Participants willtake blinded investigational product(IP) once daily
  Arms: BHV-7000 75 mg Part B
Drug: Placebo — Matching placebo taken once daily
  Arms: Placebo Part B

SUMMARY:
The purpose of this study is to determine whether BHV-7000 is effective in the treatment of refractory focal epilepsy.

DETAILED DESCRIPTION:
This study has two parts, Part A and Part B. Part A is randomized 1:1:1 25 mg of BHV-7000, 50 mg of BHV-7000 or matching placebo. Part B is randomized 1:1 75mg BHV-7000 or matching placebo. Part B will start after Part A.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and Female participants 18 to 75 years of age at time of consent.
2. Diagnosis of Focal Onset Epilepsy at least 1 year prior to screening visit defined by 2017 International League Against Epilepsy (ILAE) Classification and based on requirements of Epilepsy Adjudication criteria.

   a. Focal seizures i. Focal aware seizures with clinically observable signs and/or symptoms ii. Focal impaired awareness seizures iii. Focal to bilateral tonic-clonic seizures
3. Subject meets the 2009 ILAE definition of drug resistant epilepsy, failure of adequate trials of two tolerated and appropriately chosen and used anti-seizure medication (ASM) schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom.
4. Ability to keep accurate seizure diaries
5. Current treatment with at least 1 and up to 3 ASMs and 4 epilepsy treatments in total

Key Exclusion Criteria:

1. History of status epilepticus (convulsive status epilepticus for > 5 minutes or focal status epilepticus with impaired consciousness for > 10 minutes) within the last 6 months prior to screening visit that is not consistent with the subject's habitual seizure.
2. History of repetitive/cluster seizures (where individual seizures cannot be counted) within the last 6 months prior to screening visit and during observation phase.
3. Resection neurosurgery for seizures <4 months prior to the screening visit.
4. Radiosurgery performed <2 years prior to the screening visit.
5. Subjects with only focal aware nonmotor seizures which involve subjective sensory or psychic phenomena only, without impairment of consciousness or awareness (formally called simple partial seizures), with or without ictal EEG correlation with clinical symptoms.
6. Any condition that would interfere with the subject's ability to comply with study instructions, place the subject at unacceptable risk, and/or confound the interpretation of safety or efficacy data from the study, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part B: Change from Baseline in 28-day average seizure frequency | Baseline, Week 8 to Week 20 of Part B
  To compare the efficacy of each of 2 doses of BHV-7000 to placebo as an adjunctive therapy for refractory focal onset epilepsy as measured by the change from OP (observational phase) in 28-day average seizure frequency. The primary objective will be measured by comparing the observation phase (8 weeks) to the 12-week double-blind treatment phase.
Part A: Number of Participants With Deaths, Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and moderate or severe AEs | Week 8 to Week 20 of Part A
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with deaths, SAEs, AEs leading to discontinuation, and moderate and severe AEs.
Part A: Number of Participants With Clinically Significant Laboratory Abnormalities | Week 8 to Week 20 of Part A
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 and 4 laboratory abnormalities.

SECONDARY OUTCOMES:
Part B: Percentage of Participants with at at least 50% reduction in seizure frequency per month | Baseline, Week 8 to Week 20 of Part B
  To compare the efficacy of 2 dose strengths of BHV-7000 to placebo as adjunctive therapy for refractory focal onset epilepsy as measured by the proportion of subjects that have at least a 50% reduction in seizures per month (28 days). This objective will be measured by comparing the proportion of subjects with at least a 50% reduction in 28-day average seizure frequency over the course of the 12 week double-blind phase to the observation phase.
Part B: Change from Baseline in 28-day average seizure frequency during first month of treatment | Baseline, Week 8 to Week 12 of Part B
  To compare the efficacy of BHV-7000 to placebo during the first month of treatment. This objective will be measured by the change in log-transformed 28-day adjusted seizure frequency from observation phase over the first month of the double blind phase.
Part B: Percentage of Participants with at at least 75% reduction in seizure frequency per month | Baseline, Week 8 to Week 20 of Part B
  To compare the efficacy of BHV-7000 to placebo as measured by the proportion of subjects that have at least a 75% reduction in seizures per month (28 days). This objective will be measured by comparing the proportion of subjects with at least a 75% reduction in 28-day average seizure frequency over the course of the double-blind phase compared to the observation phase.
Part B: Percentage of Participants with seizure freedom during DB Phase | Week 8 to Week 20 of Part B
  To compare the efficacy of BHV-7000 to placebo on seizure freedom (100% seizure reduction during the DB phase). This objective will be measured by proportion of subjects that are seizure free during the double-blind phase.
Part B: Change from baseline in 7-day adjusted seizure frequency during first week of treatment | Baseline, Week 8 to Week 9 of Part B
  To compare the efficacy of BHV-7000 to placebo during the first week of treatment. This objective will be measured by the change in log-transformed 7-day adjusted seizure frequency from observation phase over the first week of the double-blind phase.
Part B: Change from baseline in Patient Global Impression of Change (PGI-C) | Baseline, Week 20 of Part B
  To compare the efficacy of BHV-7000 to placebo on the patient global impression of change (PGI-C). This objective will be measured by proportion of subjects at week 12 of double-blind treatment phase with a PGI-C response of "minimally improved", "much improved" or "very much improved". This scale is a 7-point Likert scale with response options of:
  (1) "very much improved" , (2) "much improved", (3) "minimally improved", (4) "no change", (5) "minimally worse", (6) "much worse", (7) and "very much worse"
Part B: Number of Participants With Deaths, Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and moderate or severe AEs | Week 8 to Week 20 of Part B
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with deaths, SAEs, AEs leading to discontinuation, and moderate and severe AEs.
Part B: Number of Participants With Clinically Significant Laboratory Abnormalities | Week 8 to Week 20 of Part B
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 and 4 laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (124):
- United States (61):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - WRN, Rogers, Arkansas
  - University of California San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford Health Care, Palo Alto, California
  - Profound Research LLC, Pasadena, California
  - University of Colorado Anschultz Medical Campus, Aurora, Colorado
  - Yale School of Medicine - Yale-New Haven Hospital, New Haven, Connecticut
  - EZR Research LLC, Boca Raton, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - University of Florida (Jacksonville), Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Floridian Research Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Santos Research Center, Tampa, Florida
  - Encore Medical Research of Weston LLC., Weston, Florida
  - Pediatrix Medical Group of Florida, Winter Park, Florida
  - Augusta University, Augusta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Revive Research Institute, Inc., Elgin, Illinois
  - Accellacare, Ames, Iowa
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - MAESC, Bethesda, Maryland
  - Javara, Silver Spring, Maryland
  - Revive Research Institute, Inc., Rochester Hills, Michigan
  - Minnesota Epilepsy Group, P.A., Roseville, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NEREG, Hackensack, New Jersey
  - Inst of Neurology, Livingston, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - BCHP, Hawthorne, New York
  - Northwell Health, New York, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Five Towns Neuroscience Research, Woodmere, New York
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Accellacare, Mooresville, North Carolina
  - Wake Forest Baptist, Winston-Salem, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - OSU, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Clinical Research Solutions LLC, Cypress, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Tarrant Neurology Consultants, Fort Worth, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Road Runner Research, Ltd, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - UVM MC, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Henrico Doctors Neurology Associates, LLC, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
- Argentina (10):
  - STAT Research S.A., Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital General de Agudos Dr. José María Ramos Mejia, Balvanera, Ciudad Autónoma de BuenosAires
  - Centro de Educación Médica e Investigaciones Clínicas Norberto Quirno CEMIC-Elías Galván 4102, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital Británico de Buenos Aires, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Investigaciones Sanatorio Del Sur, San Miguel de Tucumán, Tucumán Province
  - Sanatorio de la Trinidad - Mitre, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Fundación Para La Lucha Contra Las Enfermedades Neurológicas de La Infancia - FLENI, Buenos Aires
  - Instituto Privado Kremer, Córdoba
  - Conci Carpinella - Santa Rosa N° 748, Córdoba
- Austria (4):
  - Kepler Universitätsklinikum Linz - Med Campus III, Linz, Upper Austria
  - Christian Doppler-Klinik - Universitätsklinikum der PMU, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
- Belgium (5):
  - UZ Antwerpen, Edegem, Antwerpen
  - Hôpital Erasme, Anderlecht, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - CHU UCL Namur - Site Godinne, Yvoir, Namur
  - UZ Gent, Ghent, Oost-Vlaanderen
- Chile (5):
  - Centro de especialidades médicas Vanguardia, Temuco, Región de la Araucanía
  - Instituto Neurologico Thalamus, Viña del Mar, Región de Valparaíso
  - Hospital Padre Hurtado, Santiago, Región-MetropolitanadeSantiago
  - BIOCINETIC Ltda, Santiago, Región-MetropolitanadeSantiago
  - Centro de Investigacion Clinica UC, Santiago, Región-MetropolitanadeSantiago
- Croatia (3):
  - Clinical Hospital Sveti duh, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre Milosrdnice - Vinogradska cesta 29, Zagreb, City of Zagreb
  - Clinical Hospital Center Rijeka - PPDS, Rijeka
- Czechia (2):
  - Fakultni nemocnice v Motole, Prague, Praha, Hlavní Mesto
  - Fakultni nemocnice u sv. Anny v Brne, Brno, South Moravian
- France (9):
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg, Bas-Rhin
  - CHU Dijon Bourgogne, Dijon, Côte-d'Or
  - CHU de Toulouse-Hôpital Pierre-Paul Riquet-Site de Purpan, Toulouse, Haute-Garonne
  - CHU de Montpellier- Hôpital Gui De Chauliac, Montpellier, Hérault
  - CHRU de Tours - Hôpital Bretonneau, Tours, Indre-et-Loire
  - CHRU Nancy, Nancy, Meurthe-et-Moselle
  - CHU de Lille - Hopital Claude Huriez, Lille, Nord
  - Hospices Civils de Lyon - 59 Bd Pinel, Lyon, Rhône
  - Hôpital Pontchaillou, Rennes
- Hungary (4):
  - Pécsi Tudományegyetem Klinikai Kozpont -Ret u., Pécs, Baranya
  - Debreceni Egyetem Klinikai Kozpont Kenezy Gyula Campus, Debrecen, Hajdú-Bihar
  - Budapesti Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - SE INK Juhasz Pal Epilepszia Központ, Budapest
- Netherlands (3):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Stichting Epilepsie Instellingen Nederland - Heemstede, Heemstede, North Holland
  - Stichting Epilepsie Instellingen Nederland - Dokter Denekampweg 20, Zwolle, Overijssel
- Poland (14):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Przychodnia VISTAMED, Wroclaw, Lower Silesian Voivodeship
  - Clinical Best Solutions - Lublin, Lublin, Lublin Voivodeship
  - NZOZ IGNIS dr med. Alicja Lobinska, Świdnik, Lublin Voivodeship
  - Twoja Przychodnia Nowosolskie Centrum Medyczne sp. z o.o, Nowa Sól, Lubusz Voivodeship
  - Santa Familia PTG Lodz, Lodz, Lódzkie
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - Neurosphera SP. Z O.O, Warsaw, Masovian Voivodeship
  - Instytut Psychiatrii i Neurologii, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o. - ul. Nowe Ogrody 1-6, Gdansk
  - Novo-Med Zielinski i wsp. Sp.J. - ul. Brynowska 44, Katowice
  - Pratia MCM Kraków, Krakow
  - LANDA Specjalistyczne Gabinety Lekarskie, Krakow
- University Clinical Centre Maribor, Maribor, Slovenia
- South Africa (2):
  - InnoMed Clinical Trial Centre, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
- Klinik Lengg AG, Zurich, Zürich (de), Switzerland